CLINICAL TRIAL: NCT02746874
Title: Does Radiofrequency Ablation of the Articular Nerves of the Knee Prior to Total Knee Replacement Improve Pain Outcomes? A Prospective Randomized Sham-Control Trial With 6 Month Follow Up
Brief Title: Does Radiofrequency Ablation of the Articular Nerves of the Knee Prior to Total Knee Replacement Improve Pain Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Associate Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00200439
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Total Knee Replacement, Replacement of the knee joint,
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Group (Active Comparator): Radiofrequency ablation procedure of the three articular branches of the knee joint. The targets will be thermally lesioned for 2 minutes 30 seconds thereby causing neurolysis.
  Interventions: Procedure: Radiofrequency Ablation (RFA)
- Placebo Group (Sham Comparator): Simulated Radiofrequency Ablation procedure of the three articular branches of the knee joint.The targets will be not be thermally lesioned for 2 minutes 30 seconds therefore not causing neurolysis.
  Interventions: Procedure: Simulated Radiofrequency Ablation (RFA)

INTERVENTIONS:
Procedure: Radiofrequency Ablation (RFA) — The radiofrequency generator which will be turned on but will not be in the patient's view. The skin overlying the target sites identified with image guidance will be numb using lidocaine 1%. A needle will be placed through the skin to be optimally positioned according to the three targets. Sensory and motor testing will be performed to confirm appropriate placement. Lidocaine 2% 1-2cc will be injected prior to lesioning.
  Arms: Active Group
Procedure: Simulated Radiofrequency Ablation (RFA) — The radiofrequency generator which will be turned on but will not be in the patient's view. The skin overlying the target sites identified with image guidance will be numb using lidocaine 1%. A needle will be placed through the skin to be optimally positioned according to the three targets. Sensory and motor testing will be performed to confirm appropriate placement. Lidocaine 2% 1-2cc will be injected. A simulate sham lesion will be performed at each target site.
  Arms: Placebo Group

SUMMARY:
More than 300,000 total knee joint replacement surgeries are performed per year in the United States and safe, effective management of post-operative pain in these patients, often elderly, deconditioned, obese, or with co-morbid diseases like sleep apnea, can be challenging and often require a multidisciplinary, multimodal approach. Opiates have been a mainstay of treatment in the post-operative period with varying degrees of success and complications. Inadequately controlled postoperative pain is not uncommon. Poorly controlled pain inhibits early mobilization and hinders post-operative physical therapy.

A new paradigm for treating post-operative pain following total knee replacement may be the use of cooled radiofrequency ablation (C-RFA) of the articular sensory nerve supply of the knee capsule prior to surgery, to desensitize the knee by blocking sensory afferents to the anterior capsule and thereby decrease post-operative pain. There are several publications that have demonstrated the use of RFA in patients with chronic knee pain from osteoarthritis however the use of RFA in the preoperative management of pain in patients undergoing total knee joint replacement has not been investigated.

The aim of this study is to determine if patients undergoing unilateral total knee replacement obtain any post-operative pain relieving benefits from C-RFA of the articular sensory nerve supply when performed prior to surgery, as compared to sham controls who receive only local anesthetic injections of these same nerves without the benefit of ablation treatment.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee scheduled to undergo their first unilateral knee joint replacement
* willingness to undergo fluoroscopy-guided C-RFA or sham treatment

Exclusion Criteria:

* pregnancy,
* severe cardiac/pulmonary compromise,
* acute illness/infection,
* coagulopathy
* bleeding disorder,
* allergic reactions,
* contraindications to a local anesthetic

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Anesthesiology Pain Medicine Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walega D, McCormick Z, Manning D, Avram M. Radiofrequency ablation of genicular nerves prior to total knee replacement has no effect on postoperative pain outcomes: a prospective randomized sham-controlled trial with 6-month follow-up. Reg Anesth Pain Med. 2019 Apr 25:rapm-2018-100094. doi: 10.1136/rapm-2018-100094. Online ahead of print. PMID 31023931

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Group | Placebo Group
Started | 35 | 35
Completed | 35 | 32
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Surgery Date Changed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Placebo Group | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Continuous [Median (Standard Deviation); unit: Years] | 66 (7) | 66 (9) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 32 | 28 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 27 | 20 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 35 | 32 | 67
Operative site [Count of Participants; unit: Participants]
  Left Side | 19 | 14 | 33
  Right Side | 16 | 18 | 34
BMI (kg/m^2) [Median (Standard Deviation); unit: BMI (kg/m^2)] — Body mass index (BMI) index is a value derived from the mass (weight) and height.BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2
  BMI (kg/m^2) | 32.0 (5.4) | 30.5 (5.3) | 31 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption After Surgery
Description: Pain medication will be calculated into oral morphine equivalents (ME) for the first 48 hours after surgery. Morphine equivalents determine a patient's cumulative intake of any drugs in the opioid class.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: Morphine Equivalents (ME)
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
Morphine Equivalents (ME) | 192 [105 to 274] | 144 [112 to 314]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .978, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Oral Morphine Equivalent Milligrams at Baseline.
Description: The total morphine equivalent (milligrams) reported by the subject at baseline.
Time Frame: Pre operative
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
milligrams | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Oral Morphine Equivalents at Baseline Compared to 48 Hours Post-operative.
Description: Total oral morphine equivalents at baseline compared to oral morphine equivalents at 48 hours post-operative.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: Morphine Equivalents (ME)
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
Morphine Equivalents (ME) | -187 [-233 to -148] | -191 [-254 to -133]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .978, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Medication Quantification Scale III (MQSIII) Score 48 Hours Post-operative.
Description: Medication Quantification Scale III (MQSIII) is a method of quantifying different pain drug regimens by evaluating the use of 22 distinct drug classes (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs], antidepressants, benzodiazepines, opiates). A single value is calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed. The score is calculated for a given pharmacologic class by taking its detriment weight, as determined by the physician, multiplied by a score given for dosage. The scores for each pharmacologic class prescribed to a patient are then summed to determine the overall score of a given pain medication regimen. The scale ranges from (0 low (good) 500 high (poor).
Time Frame: 48 hours
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
score on a scale | 33 (8) | 35 (7)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .371, t-test, 2 sided

5. Secondary Outcome: Number of Stairs Climbed on Post-operative Day 2.
Description: Number of stairs climbed on post-operative day 2 prior to discharge from the hospital.
Time Frame: Post operative day 2
Measure: Mean (Standard Deviation); unit: stairs
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
stairs | 7 (4) | 8 (5)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .325, t-test, 2 sided

6. Secondary Outcome: Distance Walked on Post-operative Day 2.
Description: Distance in feet walked on post-operative day 2 prior to discharge from the hospital.
Time Frame: Post operative day 2
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
feet | 216 (134) | 232 (115)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .466, t-test, 2 sided

7. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score 6 Months Post Operative
Description: Western Ontario and McMaster Universities Arthritis Index (WOMAC) score 6 months post operative. The WOMAC score is a survey comprised of 24 items divided into three subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). Subjects are asked a range of questions about their ability to carry out daily activities such as using the stairs, rising from sitting, lying in bed and conducting light or heavy domestic duties. Items are scored on a scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). Values are summed up for a combined WOMAC score of 0 (low) to 96 (high) Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitation.
Time Frame: 6 months post operative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 35 | 32
score on a scale | 8 [4 to 22] | 9 [2 to 14]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .368, Wilcoxon (Mann-Whitney)

8. Post Hoc Outcome: Medication Quantification Scale Version III (MSQVIII) at Baseline in Patients With Hospital Anxiety and Depression Scores of Less Than 11.
Description: Medication Quantification Scale Version III (MQSVIII) is a single value calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed. The score is calculated for a given pharmacologic class by taking its detriment weight, as determined by the physician, multiplied by a score given for dosage. The scores for each pharmacologic class prescribed to a patient are then summed to determine the overall score of a given pain medication regimen at baseline in patients (the scale ranges from (0 low (good) 500 high) with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 29
score on a scale | 6.5 [3 to 10] | 4 [2 to 10]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .509, Wilcoxon (Mann-Whitney)

9. Post Hoc Outcome: Medication Quantification Scale Version III (MSQVIII) at 48 Hours in Patients With Hospital Anxiety and Depression Scores of Less Than 11.
Description: Medication Quantification Scale Version III (MQSVIII) is a single value calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed. The score is calculated for a given pharmacologic class by taking its detriment weight, as determined by the physician, multiplied by a score given for dosage. The scores for each pharmacologic class prescribed to a patient are then summed to determine the overall score of a given pain medication regimen score on a scale of 0 good-500 poor at baseline in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 27
score on a scale | 33.5 [28 to 37] | 34 [30 to 38]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .593, Wilcoxon (Mann-Whitney)

10. Post Hoc Outcome: Medication Quantification Scale Version III (MSQVIII) at 1 Month in Patients With Hospital Anxiety and Depression Scores of Less Than 11.
Description: Medication Quantification Scale Version III (MQSVIII) is a single value calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed. The score is calculated for a given pharmacologic class by taking its detriment weight, as determined by the physician, multiplied by a score given for dosage. The scores for each pharmacologic class prescribed to a patient are then summed to determine the overall score of a given pain medication regimen (score on a scale 0 good-500 poor) at baseline in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 27
score on a scale | 7 [3 to 7.5] | 5 [0 to 9]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = 0.687, Wilcoxon (Mann-Whitney)

11. Post Hoc Outcome: Medication Quantification Scale Version III (MSQVIII) at 6 Months in Patients With Hospital Anxiety and Depression Scores of Less Than 11.
Description: Medication Quantification Scale Version III (MQSVIII) is a single value calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed. The score is calculated for a given pharmacologic class by taking its detriment weight, as determined by the physician, multiplied by a score given for dosage. The scores for each pharmacologic class prescribed to a patient are then summed to determine the overall score of a given pain medication regimen (the scale ranges from (0 low (good) 500 high) at baseline in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 29 | 27
score on a scale | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .813, Wilcoxon (Mann-Whitney)

12. Post Hoc Outcome: Medication Quantification Scale Version III (MSQVIII) at 3 Months in Patients With Hospital Anxiety and Depression Scores of Less Than 11.
Description: as for outcome 10
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 27
score on a scale | 0 [0 to 4.5] | 0 [0 to 6]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .687, Wilcoxon (Mann-Whitney)

13. Post Hoc Outcome: Total Oral Morphine Equivalents in Milligrams at Baseline in Patients With Hospital Anxiety and Depression Scores (HADS) of Less Than 11.
Description: Total oral morphine equivalents in milligrams at baseline in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 29
milligrams | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = 0.840, Wilcoxon (Mann-Whitney)

14. Post Hoc Outcome: Total Oral Morphine Equivalents in Milligrams at 48 Hours in Patients With Hospital Anxiety and Depression Scores (HADS) of Less Than 11.
Description: Total oral morphine equivalents in milligrams at 48 hours in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 29
milligrams | 178.5 [92.5 to 267] | 138 [110 to 328]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .913, Wilcoxon (Mann-Whitney)

15. Post Hoc Outcome: Total Oral Morphine Equivalents in Milligrams at 1 Month in Patients With Hospital Anxiety and Depression Scores (HADS) of Less Than 11.
Description: Total oral morphine equivalents in milligrams at 1 month in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 1 month post operative
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 27
milligrams | 10 [1 to 20] | 5 [0 to 10]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = 0.301, Wilcoxon (Mann-Whitney)

16. Post Hoc Outcome: Total Oral Morphine Equivalents in Milligrams at 3 Months in Patients With Hospital Anxiety and Depression Scores (HADS) of Less Than 11.
Description: Total oral morphine equivalents in milligrams at 3 months in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 3 month post operative
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 27
milligrams | 0 [0 to 4] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = 0.826, Wilcoxon (Mann-Whitney)

17. Post Hoc Outcome: Total Oral Morphine Equivalents in Milligrams at 6 Months in Patients With Hospital Anxiety and Depression Scores (HADS) of Less Than 11.
Description: Total oral morphine equivalents in milligrams at 6 months in patients with Hospital Anxiety and Depression Scores (HADS) of less than 11.The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 6 month post operative
Measure: Median (Inter-Quartile Range); unit: Milligrams
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 29 | 27
Milligrams | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .813, Wilcoxon (Mann-Whitney)

18. Post Hoc Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at Baseline in Patients With Hospital Anxiety and Depression Scale (HADS) Scores of Less Than 11.
Description: WOMAC score at baseline in patients with Hospital Anxiety and Depression Scale (HADS) Scores of less than 11.The WOMAC score is a survey comprised of 24 items divided into three subscales:Pain (5 items), stiffness (2 items), and physical function (17 items). Subjects are asked a range of questions about their ability to carry out daily activities such as using the stairs, rising from sitting, lying in bed and conducting light or heavy domestic duties. Items are scored on a scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). Summed for a combined WOMAC score of 0 (low) to 96 (high) Higher scores indicate worse pain, stiffness, and functional limitation. The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression.The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 29
score on a scale | 39.5 [32.5 to 52] | 40 [22 to 48]

19. Post Hoc Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 1 Month in Patients With Hospital Anxiety and Depression Scale (HADS) Scores of Less Than 11.
Description: WOMAC score at 1 month in patients with Hospital Anxiety and Depression Scale (HADS) Scores of less than 11.The WOMAC score is a survey comprised of 24 items divided into three subscales:Pain (5 items), stiffness (2 items), and physical function (17 items). Subjects are asked a range of questions about their ability to carry out daily activities such as using the stairs, rising from sitting, lying in bed and conducting light or heavy domestic duties. Items are scored on a scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). Summed for a combined WOMAC score of 0 (low) to 96 (high) Higher scores indicate worse pain, stiffness, and functional limitation. The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression.The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 1 month post operative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 32 | 27
score on a scale | 21 [14 to 28] | 13 [8 to 22]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .047, Wilcoxon (Mann-Whitney)

20. Post Hoc Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 3 Month in Patients With Hospital Anxiety and Depression Scale (HADS) Scores of Less Than 11.
Description: WOMAC score at 3 months in patients with Hospital Anxiety and Depression Scale (HADS) Scores of less than 11.The WOMAC score is a survey comprised of 24 items divided into three subscales:Pain (5 items), stiffness (2 items), and physical function (17 items). Subjects are asked a range of questions about their ability to carry out daily activities such as using the stairs, rising from sitting, lying in bed and conducting light or heavy domestic duties. Items are scored on a scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). Summed for a combined WOMAC score of 0 (low) to 96 (high) Higher scores indicate worse pain, stiffness, and functional limitation. The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression.The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 3 month post operative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 29 | 27
score on a scale | 11.5 [6 to 23.5] | 8 [2 to 17]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .115, Wilcoxon (Mann-Whitney)

21. Post Hoc Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 6 Month in Patients With Hospital Anxiety and Depression Scale (HADS) Scores of Less Than 11.
Description: WOMAC score at 6 months in patients with Hospital Anxiety and Depression Scale (HADS) Scores of less than 11.The WOMAC score is a survey comprised of 24 items divided into three subscales:Pain (5 items), stiffness (2 items), and physical function (17 items). Subjects are asked a range of questions about their ability to carry out daily activities such as using the stairs, rising from sitting, lying in bed and conducting light or heavy domestic duties. Items are scored on a scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). Summed for a combined WOMAC score of 0 (low) to 96 (high) Higher scores indicate worse pain, stiffness, and functional limitation. The Hospital Anxiety and Depression Scores (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression.The questionnaire is scored from 0-3 and this means that a person can score between 0 (low) and 21 (high) for either anxiety or depression.
Time Frame: 6 month post operative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 29 | 27
score on a scale | 9 [4 to 20] | 9 [1 to 14]
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority; p = .349, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Collection of adverse events 48 hours after total knee arthroplasty.
Arm/Group | Active Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 8/35 | 9/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Group (N=35) | Placebo Group (N=32)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9)
Puritis (Skin and subcutaneous tissue disorders) | 8 (8) | 9 (9) — Puritis experienced up to 48 hours after surgery.

LIMITATIONS AND CAVEATS:
During the study 2016-2018 there was increased patient and physician awareness of opioid abuse epidemic in the US. Fear of opioid addiction and increased pressure on physician may have influenced post operative opioid use and primary outcome

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT02746874/Prot_SAP_000.pdf